CLINICAL TRIAL: NCT03729232
Title: Japanese Catheter Ablation Registry
Acronym: J-AB
Status: Recruiting | Type: Observational
Sponsor: National Cerebral and Cardiovascular Center, Japan (Other)
Responsible Party: Principal Investigator, Kengo Kusano, Director of Cardiovascular Medicine, National Cerebral and Cardiovascular Center, National Cerebral and Cardiovascular Center, Japan
Other Study IDs: M28-114; UMIN000028288 (Other: UMIN-CTR)
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Catheter Ablation; Cardiac Arrhythmias
Keywords: Catheter Ablation; Cardiac Arrhythmias; Registry; Complication; REDCap
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Japanese Cather Ablation (J-AB) Registry is a voluntary nationwide registry, performed by Japanese Heart Rhythm Society, collaborated with the National Cerebral and Cardiovascular Center. The objectives of this registry are to observe and describe developments in the catheter ablation treatment of arrhythmia in Japan and to provide reliable information on the type of activity performed and the facilities available in Japanese arrhythmia units.

DETAILED DESCRIPTION:
Japanese Cather Ablation (J-AB) Registry is a nationwide, multicenter, observational registry, performed by Japanese Heart Rhythm Society, collaborated with National Cerebral and Cardiovascular Center.

This study is a voluntary nationwide registry and data are collected prospectively using a Research Electronic Data Capture (REDCap) system. Detailed data collection including antiarrhythmic medication is also performed at every September. The acute success rate at discharge and the complications associated with ablation procedure will be collected in all cases. Major bleeding events are defined according to Bleeding Academic Research Consortium criteria. Based on the provided information, the annual incidence and predictive factors for outcome will be investigated by the event assessment committee.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with catheter ablation in Japan

Exclusion Criteria:

* Patients who refused to consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inpatients
Sampling Method: Non-Probability Sample
Enrollment: 400000 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with recurrence of targeted arrhythmia | Through discharge from hospital, approximately up to 1 weeks

SECONDARY OUTCOMES:
Number of deaths | Through discharge from hospital, approximately up to 1 weeks
  All-cause death, cardiovascular death, and procedure-related death
Number of patients with treatment-related complications | 3 months
  Bleeding events, embolic events, other all complications. Major bleeding events are defined according to Bleeding Academic Research Consortium criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Teiichi Yamane, MD, PhD, Principal Investigator — The Jikei University School of Medicine; Kengo Kusano, MD, PhD, Principal Investigator — National Cerebral and Cardiovascular Center, Japan
Locations (1):
- National Cerebral and Cardiovascular Center, Suita, Osaka, Japan

REFERENCES:
- [Derived] Matsuda Y, Masuda M, Kanaoka K, Mano T, Inoue K, Yamashita S, Iwasaki YK, Nakamura K, Nagashima K, Miyamoto K, Satomi K, Takatsuki S, Kusano K, Yamane T, Shimizu W. Real-World Outcomes of Repeat Ablation Strategies for Atrial Fibrillation: Insights From the Japanese Catheter Ablation Registry. J Arrhythm. 2025 Sep 22;41(5):e70200. doi: 10.1002/joa3.70200. eCollection 2025 Oct. PMID 40995616
- [Derived] Goto K, Miyazaki S, Tonegawa-Kuji R, Kanaoka K, Yamashita S, Sasano T, Iwanaga Y, Nakai M, Inoue K, Iwasaki YK, Nagashima K, Nakamura K, Masuda M, Miyamaoto K, Satomi K, Takatsuki S, Kusano K, Yamane T, Shimizu W. Efficacy and Safety of Second Sessions of Catheter Ablation for Idiopathic Premature Ventricular Contractions: From the Nationwide Japan Catheter Ablation Registry. J Arrhythm. 2025 Aug 25;41(4):e70181. doi: 10.1002/joa3.70181. eCollection 2025 Aug. PMID 40861252
- [Derived] Oikawa J, Fukaya H, Kanaoka K, Niwano S, Miyamoto K, Iwanaga Y, Iwasaki YK, Nagashima K, Masuda M, Yamashita S, Nakamura K, Satomi K, Takatsuki S, Inoue K, Kusano K, Yamane T, Tada H, Shimizu W. Efficacy and safety of catheter ablation for paroxysmal atrial fibrillation: A comparison of first-line vs second-line therapy. Heart Rhythm. 2025 Jul 24:S1547-5271(25)02711-0. doi: 10.1016/j.hrthm.2025.07.030. Online ahead of print. PMID 40714332